CLINICAL TRIAL: NCT06000098
Title: Effect of Console Time on the Development of Acute Kidney Injury in Robotic-assisted Laparoscopic Prostatectomy
Brief Title: Consol Time and Acute Kidney Injury in Robotic-assisted Prostatectomy
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: ATADEK 2021-01/2
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Acute Kidney Injury; Hemodynamic Instability
Keywords: Robotic-assisted laparoscopic prostatectomy; Acute kidney injury; Restrictive fluid therapy; Pressure recording analytical method
MeSH Terms: conditions — Acute Kidney Injury | interventions — Head-Down Tilt

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing robotic-assisted laparoscopic prostatectomy in deep Trendelenburg position.: Patients with ASA( American Society of Anesthesiologists) physical status 1-3 who underwent robotic-assisted laparoscopic prostatectomy in deep Trendelenburg position with restrictive fluid therapy
  Interventions: Other: Restrictive fluid therapy

INTERVENTIONS:
Other: Restrictive fluid therapy — 0,5 ml/hour fluid administration during prostatic anastomosis.
  After general anesthesia induction, the patients were placed in the deep Trendelenburg position (at least 25°-45° upside down).
  Other Names: Trendelenburg position.

SUMMARY:
Robotic-assisted laparoscopic prostatectomy (RALP) is the gold standard surgical technique in prostate surgery. Many Robotic-laparoscopic surgical techniques also require the intraoperative deep Trendelenburg position and intravenous fluid restriction during surgery. However, the possible side effects of the deep Trendelenburg's position and the fluid restriction on the cardiovascular and renal systems during surgery are unknown. Although the Trendelenburg position is a life-saving maneuver in hypovolemic patients, it also carries undesirable risks. Long console time may contribute to the development of acute kidney injury (AKI) by prolonging the Trendelenburg time and the fluid-restricted time. In this study, investigators aimed to demonstrate the effect of console time on the development of AKI. Investigators also aimed to determine the hemodynamic risk factors that cause the development of AKI in patients monitored with the pressure Recording Analytical Method (PRAM).

DETAILED DESCRIPTION:
Although open surgery has been used for a long time in the treatment of prostate diseases, robotic-assisted laparoscopic prostatectomy (RALP) has become more common in the last 20 years. The excellence in results has made the use of the robot the gold standard in prostate surgery. However, the presence of two critical factors during RALP surgery still bothers clinicians. The first of these is severe fluid restriction and the other is the deep Trendelenburg position and pneumoperitoneum. The prolongation of the robotic console time also causes the prolongation of fluid restriction and Trendelenburg time. This combination may cause significant pathophysiological changes in both the renal and cardiac systems and may lead to postoperative acute renal injury (AKI). AKI is a serious clinical complication with increasing incidence and is associated with adverse short-term and long-term outcomes worldwide, resulting in a large healthcare burden. Intraoperative advanced monitoring techniques can contribute to the prevention of renal damage that may occur by providing early recognition of these pathophysiological changes occurring in the renal and cardiac systems.

The aim of our study was to determine the effect of console duration on the incidence of AKI after RALP which was managed using intraoperative advanced monitoring techniques (pressure recording analytical method-PRAM). In addition, this study aimed to evaluate the ability of changes in hemodynamic parameters to predict the development of AKI in RALP patients who underwent restrictive fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society Of Anesthesiology physical status 1-3
* Underwent Robotic-assisted laparoscopic prostatectomy
* Underwent restrictive fluid therapy during the console period

Exclusion Criteria:

* Under 18 years of age
* Arrhythmia (atrial fibrillation, frequent premature beat)
* History of myocardial infarction in the last 3 months
* Heart failure
* Severe pre-existing lung disease
* Severe valvular heart disease
* Chronic renal disease on dialysis,

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with ASA (American Society Of Anesthesiology) physical status 1-3 who underwent RALP with restrictive fluid therapy during console period
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Console time was measured for evaluating the effect of restrictive fluid therapy and prostatic urethra anastomosis time on the development of acute kidney injury. | The duration of the measurement was defined as during the surgery.
  Console time ( minute) indicates the restrictive fluid therapy time, prostatic resection, and prostatic urethra anastomosis time.

SECONDARY OUTCOMES:
Stroke volume variation (SVV) was measured for evaluation of volume status | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Stroke volume variation (SVV,%), was monitored using the pressure recording analytic method. SVV is a parameter used to asses cardiac preload and fluid responsiveness.
Pulse pressure variation (PPV) was measured for evaluation of volume status | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Pulse pressure variation (PPV,%) was monitored using the pressure recording analytic method. PPV is a parameter used to asses cardiac preload and fluid responsiveness
Cardiac power output (CPO) was measured for evaluation of cardiac power reserve | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Cardiac power output (CPO, Watt) was monitored using the pressure recording analytic method. CPO is a parameter used to asses cardiac reserve
Cardiac index (CI) was measured for evaluating cardiac flow | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Cardiac index (CI, L/min/m2), was monitored using the pressure recording analytic method. CI is a parameter used to asses cardiac stroke volume.
Dp/Dt was measured to assess cardiac systolic function | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Dp/Dt(mmHg/msn), was monitored using the pressure recording analytic method. Dp/Dt is a parameter used to asses cardiac contractility.
Systolic arterial pressure (SAP) was measured for evaluating perfusion pressure | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Systolic arterial pressure (SAP- mm/Hg) was monitored using the pressure recording analytic method. SAP is a parameter used to assess the pressure of the arterial system during cardiac systole
Diastolic arterial pressure (DAP) was measured for evaluating perfusion pressure | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Diastolic arterial pressure (DAP, mm/Hg) was monitored using the pressure recording analytic method. DAP is a parameter used to assess the pressure of the arterial system during cardiac diastole
Mean arterial pressure (MAP) was measured for evaluating perfusion pressure | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Mean arterial pressure (MAP, mm/Hg) was monitored using the pressure recording analytic method. MAP is a parameter used to assess organ perfusion
Heart rate (HR) was measured for evaluating heart ritm | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Heart rate( HR, bpm) was monitored using the pressure recording analytic method. HR is a parameter used to assess the cardiac rate
Arterial elastance ( Ea) was measured for evaluation of cardiac afterload and arterial ton | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Ea ((mmHg m-2ml-1) was monitored using the pressure recording analytic method. Ea is a parameter used to assess cardiac afterload and arterial tone
The Kidney Disease: Improving Global Outcomes (KDIGO) criteria were used for the definition and staging of acute kidney injury . | The duration of the measurement was defined from the end of the surgery to the 3 days after surgery
  KDIGO criteria ( stage) classify acute kidney injury based on changes in serum creatinine levels and urine output.

CONTACTS AND LOCATIONS:
Overall Officials: Fevzi Toraman, M.D., Study Director — Acibadem Mehmet Ali Aydinlar University School of Medicine, Department of Anesthesiology
Locations (1):
- Acibadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Joo EY, Moon YJ, Yoon SH, Chin JH, Hwang JH, Kim YK. Comparison of Acute Kidney Injury After Robot-Assisted Laparoscopic Radical Prostatectomy Versus Retropubic Radical Prostatectomy: A Propensity Score Matching Analysis. Medicine (Baltimore). 2016 Feb;95(5):e2650. doi: 10.1097/MD.0000000000002650. PMID 26844486
- [Background] Sudfeld S, Leyh-Bannurah SR, Budaus L, Graefen M, Reese PC, von Breunig F, Reuter DA, Saugel B. Impact of perioperative administration of 6 % hydroxyethyl starch 130/0.4 on serum cystatin C-derived renal function after radical prostatectomy: a single-centre retrospective study. BMC Anesthesiol. 2016 Aug 30;16(1):69. doi: 10.1186/s12871-016-0236-8. PMID 27576693
- [Background] Lestar M, Gunnarsson L, Lagerstrand L, Wiklund P, Odeberg-Wernerman S. Hemodynamic perturbations during robot-assisted laparoscopic radical prostatectomy in 45 degrees Trendelenburg position. Anesth Analg. 2011 Nov;113(5):1069-75. doi: 10.1213/ANE.0b013e3182075d1f. Epub 2011 Jan 13. PMID 21233502
- [Result] Emir NS, Akyol D, Sabaz MS, Karadag S. Robotic assited perineal prostatectomy (RAPP) as a new era for anesthesiology: It's effects on hemodynamic parameters and respiratory mechanics. J Robot Surg. 2023 Jun;17(3):933-940. doi: 10.1007/s11701-022-01482-x. Epub 2022 Nov 16. PMID 36383279
- [Result] Valdivieso RF, Hueber PA, Zorn KC. Robot assisted radical prostatectomy: how I do it. Part I: Patient preparation and positioning. Can J Urol. 2013 Oct;20(5):6957-61. PMID 24128839
- [Result] Karaveli A, Kavakli AS, Cakin O, Aykal G, Yildiz A, Ates M. Comparison of plasma neutrophil gelatinase-associated lipocalin (NGAL) levels after robot-assisted laparoscopic and retropubic radical prostatectomy: an observational study. Braz J Anesthesiol. 2022 Jan-Feb;72(1):21-28. doi: 10.1016/j.bjane.2021.03.003. Epub 2021 Apr 2. PMID 33819496
- [Result] Pawlik MT, Prasser C, Zeman F, Harth M, Burger M, Denzinger S, Blecha S. Pronounced haemodynamic changes during and after robotic-assisted laparoscopic prostatectomy: a prospective observational study. BMJ Open. 2020 Oct 5;10(10):e038045. doi: 10.1136/bmjopen-2020-038045. PMID 33020097